CLINICAL TRIAL: NCT05118113
Title: Development of a Cell Culture Process for the Production of Human T-lymphocyte Precursors
Acronym: SMART101-HV1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Smart Immune SAS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SI101-HV1
Record Dates: First submitted 2021-11-05; First posted 2021-11-11 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-07

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy donors (Other)
  Interventions: Procedure: Collection of mobilized hematopoietic stem cells (apheresis products) from healthy volunteers

INTERVENTIONS:
Procedure: Collection of mobilized hematopoietic stem cells (apheresis products) from healthy volunteers — Mobilisation of hematopoietic stem cells by injection of filgrastim (authorized auxiliary medicinal product) for 4 consecutive days and leukapheresis on Day 5

SUMMARY:
The purpose of this study is to finalise the development of a process for the production of T-cell progenitor cells.

ELIGIBILITY:
Inclusion Criteria:

* Healthy donors, men aged 18 to 40 years.
* Body weight ≥ 65 kg with a body mass index (BMI) calculated by weight in kg/(height in m)² of 20 to 30 kg/m² at screening.
* Informed consent form signed and dated prior to any study-specific screening procedure.
* Health status judged by the investigator to be compatible with participation in the study based on medical history, results of physical examination, results of biological laboratory tests (cell blood count including RBC, hematocrit, hemoglobin, reticulocytes, WBC, platelet, PT, aPTT, CRP, fasting blood glucose, ionogram (Na+, K+, Cl-, HCO3-), creatinine, creatinine clearance by Cockcroft, albumin, total protein, total bilirubin, AST, ALT, ALP, GGT), vital signs measurements and 12-lead ECG. All results should be normal or, if out of range, clinically insignificant in the judgement of the investigator.
* Venous capital compatible with leukapheresis
* Have a high probability of complying with and completing the study.
* Be affiliated with a Social Security scheme

Exclusion Criteria:

* Any cardiovascular (e.g. heart failure), hepatic, renal, respiratory (e.g. asthma), gastrointestinal, endocrine (e.g. diabetes, dyslipidemia), immunological, dermatological, haematological (including hemoglobinopathy), neurological, psychiatric disorder or any history of allergy to a drug.
* State of acute illness (e.g., vomiting, fever, diarrhea) within 7 days prior to the first day of the study.
* History of drug abuse in the year preceding the first day of the study.
* History of alcoholism in the year prior to day 1 defined as consumption of more than 3 standard drinks/day (30 g/day) or 15 standard drinks/week (150 g/week) or less than two non-alcoholic days each week, or more than 5 standard drinks (50 g) on a single occasion.
* Any contra-indication to filgrastim
* Positive serological results for human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibodies, syphilis and/or human T-lymphotropic virus (HTLV).
* Positive urine drug tests (methadone, barbiturates, benzodiazepines, tricyclic antidepressants, cocaine, cannabinoids, morphine, amphetamines and methamphetamines, including 3,4-methylenedioxy-N-methylamphetamine [MDMA]).
* Laboratory workup including blood count, fasting blood glucose, blood ionogram, creatinine, AST, ALT, gamma GT, alkaline phosphatase, total bilirubin, CRP, PT, aPTT incompatible with leukapheresis protocol.
* Use of any experimental drug within 30 days prior to inclusion.
* Use of any prescription or over-the-counter medication within 5 times the elimination half-life prior to inclusion. However, any prescribed medication that may interfere with the study objectives must be discontinued for at least 30 days.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2022-04-26 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Production of cell therapy products fulfilling the required specifications | 7 days
  Production of cell therapy products fulfilling the required specifications after 7 days of CD34+ cell culture

CONTACTS AND LOCATIONS:
Overall Officials: Joe-Elie Salem, MD, PhD, Principal Investigator — CIC Paris Est, Hôpital Pitié Salpêtrière, Paris
Locations (1):
- CIC Paris Est, Hôpital Pitié Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: No